CLINICAL TRIAL: NCT07358416
Title: Determination the Safety of Disaggregant and Anticoagulant Therapy in the Development of Complications in Noncardiac Vascular Surgery.
Brief Title: Complications and Antiplatelet and Anticoagulant Therapy in Vascular Surgery.
Status: Active, not recruiting | Type: Observational
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: ComplVasc2025Retro
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Thrombosis; Bleeding; Cerebral Hypoxia During and/or Resulting From A Procedure
Keywords: Vascular surgery; Antiplatelet; Anticoagulants; complication; trombosis; bleeding
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Aspirin; Clopidogrel; Ticagrelor; Dabigatran; Rivaroxaban; apixaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Patients who did not take antiplatelet agents and anticoagulants
- Antiplatelet and anticoagulants: Patients who use antiplatelet agents and anticoagulants until the operation day
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: Ticagrelor; Drug: Dabigatran; Drug: Rivaroxaban; Drug: Apixaban; Drug: Warfarin; Drug: aspirin + clopidogrel; Drug: Aspirin + Ticagrelor; Drug: Aspirin + Apixaban; Drug: Aspirin + rivaroxaban; Drug: Clopidogrel + Apixaban; Drug: Clopidogrel + Rivaroxaban
- Discontinuation of antiplatelet and anticoagulants: Patients who discontinuate antiplatelet agents and anticoagulants until the operation day

INTERVENTIONS:
Drug: Aspirin — Patients who take aspirin until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Clopidogrel — Patients who take clopidogrel until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Ticagrelor — Patients who take ticagrelor until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Dabigatran — Patients who take dabigatran until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Rivaroxaban — Patients who take rivaroxaban until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Apixaban — Patients who take apixaban until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Warfarin — Patients who take warfarin until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: aspirin + clopidogrel — Patients who take aspirin and clopidogrel until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Aspirin + Ticagrelor — Patients who take aspirin and ticagrelor until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Aspirin + Apixaban — Patients who take aspirin and apixaban until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Aspirin + rivaroxaban — Patients who take aspirin and rivaroxaban until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Clopidogrel + Apixaban — Patients who take clopidogrel and apixaban until the operation day
  Groups: Antiplatelet and anticoagulants
Drug: Clopidogrel + Rivaroxaban — Patients who take clopidogrel and rivaroxaban until the operation day
  Groups: Antiplatelet and anticoagulants

SUMMARY:
The goal of this retrospective clinical trial is to find out association antiplatelet and anticoagulant therapy with perioperative complications in non-cardiac vascular surgery in patients . The main questions it aims to answer are:

Does the use of antiplatelet agents and anticoagulants affect the development of complications in the perioperative period during operations on the main arteries? Does discontinuing antiplatelet and anticoagulant medications affect the development of perioperative complications in major artery surgeries?? Researchers will compare with patients who didn't use antiplatelets and anticoagulant drugs to see ift he incidence of complications comparable?

This is a retrospective study based on the analysis of medical records (case histories).

ELIGIBILITY:
Inclusion Criteria:

* Patients who received surgical treatment on the main arteries.

Exclusion Criteria:

* Patients who received surgical treatment on the main veins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with surgical treatment of atherosclerotic lesions of the main arteries.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Bleeding | First 24 hours after operation
  Case of bleeding or haematoma development

SECONDARY OUTCOMES:
Trombosis | First 24 hours after operation

CONTACTS AND LOCATIONS:
Locations (1):
- NRCS Petrovsky, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes